CLINICAL TRIAL: NCT01708512
Title: Feasibility Study: Evaluation of the Ulthera® System for Lifting and Tightening of Facial and Neck Skin Laxity Using a Customized, High-Density and Vectoring Treatment Approach
Brief Title: Feasibility Study: Higher Density Ulthera® System Treatment With Vectoring for Treatment of the Face and Neck
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ulthera, Inc (Industry)
Responsible Party: Sponsor
Organization: Merz North America, Inc. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: ULT-130
Record Dates: First submitted 2012-10-15; First posted 2012-10-17 (Estimated); Last update posted 2017-11-24 (Actual); Status verified 2013-09

CONDITIONS: Skin Laxity
Keywords: Ulthera® System; Ultherapy™ Treatment; Ulthera, Inc.; Ultrasound treatment for skin tightening
MeSH Terms: conditions — Cutis Laxa

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ultherapy™ study treatment (Experimental): Each subject will receive a customized, high-density, vectored Ulthera System Treatment.
  Interventions: Device: Ulthera System Treatment

INTERVENTIONS:
Device: Ulthera System Treatment — Focused ultrasound energy delivered below the surface of the skin
  Other Names: Ultherapy™

SUMMARY:
All enrolled subject will receive one Ultherapy™ treatment. Study images will be obtained pre-treatment, immediate post-treatment, and at each study follow-up visit. Enrolled subjects will return for follow-up visits at 90 days, 180 days and 365 days post-treatment.

DETAILED DESCRIPTION:
This is a prospective, single-center clinical trial to evaluate the efficacy of the Ulthera® System to provide a customized, high-density, vectored Ultherapy™ treatment to lift and tighten the skin of the face and neck. Skin laxity changes from baseline will be assessed at study follow-up visits. Global Aesthetic Improvement Scale scores and patient satisfaction questionnaires will also be obtained.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged 25 to 60 years.
* Subject in good health.
* Skin laxity in the area(s) to be treated.
* Understands and accepts the obligation not to undergo any other procedures in the area(s) to be treated through the follow-up period.
* Willingness and ability to comply with protocol requirements, including returning for follow-up visits and abstaining from exclusionary procedures for the duration of the study.

Exclusion Criteria:

* Presence of an active systemic or local skin disease that may affect wound healing.
* Severe solar elastosis.
* Excessive subcutaneous fat in the area(s) to be treated.
* Excessive skin laxity on the area(s) to be treated.
* Significant scarring in area(s) to be treated.
* Open wounds or lesions in the area(s) to be treated.
* Severe or cystic acne on the area(s) to be treated.
* Presence of a metal stent or implant in the area(s) to be treated.
* Inability to understand the protocol or to give informed consent.
* BMI equal to and greater than 30.

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2012-04; Primary Completion 2012-12 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Improvement in overall lifting and tightening of the skin | 90 days post-treatment
  As determined by a masked, qualitative assessment of photographs at 90 days post treatment compared to baseline. The clinical response of Ulthera treatment will be assessed by comparing photographic images taken before and after the procedure.

SECONDARY OUTCOMES:
Overall aesthetic improvement | 365 days post-treatment
  Global Aesthetic Improvement Scale scores will be obtained from the Investigator and subject, assessing improvement in skin laxity based on a comparison of post-treatment photos to pre-treatment photos.

CONTACTS AND LOCATIONS:
Overall Officials: William P Werschler, MD, Principal Investigator
Locations (1):
- Premier Clinical Research, Spokane, Washington, United States

REFERENCES:
- [Derived] Werschler WP, Werschler PS. Long-term Efficacy of Micro-focused Ultrasound with Visualization for Lifting and Tightening Lax Facial and Neck Skin Using a Customized Vectoring Treatment Method. J Clin Aesthet Dermatol. 2016 Feb;9(2):27-33. PMID 27047630